CLINICAL TRIAL: NCT00197938
Title: Does the Concentration of L-Lactate in the Rectum Correlate With Mortality and Morbidity in Patients With Septic Shock?
Brief Title: Lactic Acid in the Rectum and Life-Threatening Infection
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Other Study IDs: KA 05091m
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Measurement of rectal lactic acid.

SUMMARY:
Life-threatening infection impairs bloodflow to the gut, thereby causing less delivery of oxygen. This leads to increased formation of lactic acid.

The investigators hypothesize, that the more serious the condition, the higher the concentration of lactic acid will be, thus relating to the risk of multiple organ failure or death.

ELIGIBILITY:
Inclusion Criteria:

* Fluid resuscitated septic shock < 24 h.

Exclusion Criteria:

* Septic shock > 24 h.
* Pathology in the rectum.
* Bleeding per rectum.
* Limitation of therapy.
* Where informed consent from relatives cannot be obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with early septic shock (< 24 h).
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2005-11; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Perner, MD, PhD, Study Chair — Dept. of Anaesthesia and Intensive Care, Herlev University Hospital, DK-2730 Herlev
Locations (5):
- Denmark (4):
  - Dept. of Intensive Care 4131, Rigshospitalet, Copenhagen
  - Dept. of Intensive Care, Glostrup University Hospital, Glostrup Municipality
  - Dept. of Intensive Care, Gentofte University Hospital, Hellerup
  - Dept. of Intensive Care, Herlev University Hospital, Herlev
- Dept. of Intensive Care, Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Ibsen M, Tenhunen J, Wiis J, Waldau T, Lauritsen AO, Thornberg K, Joensen H, Perner A. Lactate concentrations in the rectal lumen in patients in early septic shock. Acta Anaesthesiol Scand. 2010 Aug;54(7):827-32. doi: 10.1111/j.1399-6576.2010.02263.x. Epub 2010 Jun 15. PMID 20560883